CLINICAL TRIAL: NCT03798041
Title: Early Debridement Within 24 Hours After Surgery Compared Routine Debridement (24 Hours Later) for Wound Healing of Abdominal Incision
Brief Title: Early Debridement Within 24 Hours After Surgery for Wound Healing of Abdominal Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AFCRC2017SJ-007-1
Record Dates: First submitted 2019-01-01; First posted 2019-01-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-03

CONDITIONS: Surgical Wound
Keywords: Surgical Wound; Suture, Complication
MeSH Terms: conditions — Surgical Wound | interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debridement group (Experimental): The subjects in this group will be debrided within 24 hours after surgery.
  Interventions: Behavioral: Debridement Within 24 Hours After Surgery
- Control group (No Intervention): The subjects in this group will experience wound dressing change regularly 24 hours after surgery.

INTERVENTIONS:
Behavioral: Debridement Within 24 Hours After Surgery — Debrided within 24 hours after surgery
  Arms: Debridement group

SUMMARY:
Wound healing after surgery is a complex procedure. Liquefaction of the fat and necrosis of inactivated tissue, as well as blood clots are always accumulated mostly within 24 hours after surgery. As such, early debridement within 24 hours after surgery might improve the healing of the wounds. This study is designed to compare the impact of early debridement of the wound versus regular dressing (24 hours later) on the wound healing. 100 patients will be included in this study, and divided into 2 groups randomly. Then, the healing of the wound, stitch removal time, incidence of incision complications will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* the patient with major abdominal incision.

Exclusion Criteria:

* Pregnant woman
* Patient with diabetes
* Patient with a history of cardiovascular disease, including coronary heart disease and stroke.
* Severe lung diseases such as COPD and asthma
* Patients undergoing emergent surgery or infectious surgery
* Patients with surgical site infection or abdominal abscess
* No autonomy, inability or unwillingness to participate in follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
healing time, d (day) | From date of surgery to the date of stitches off (up to 1 month)
  since the ending of surgery to stitches off.

SECONDARY OUTCOMES:
incidence of incision complications | From the date of surgery to stitches off (up to 1 month)
  The incision complications include infection, dehiscence, fat liquefaction, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xu-Feng Zhang, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No